CLINICAL TRIAL: NCT05835986
Title: An Open-label, Multicenter, Dose Escalation, First-in-Human Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneously Administered RO7507062 in Participants With Systemic Lupus Erythematosus
Brief Title: A First-in-Human Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RO7507062 in Participants With Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BP44315; 2022-502632-39-00 (EU CTIS Number)
Record Dates: First submitted 2023-04-19; First posted 2023-04-28 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: SAD: RO7507062 (Experimental): Participants will receive RO7507062 at an assigned dose as subcutaneous (SC) injection on Day 1.
  Interventions: Drug: RO7507062; Drug: Tocilizumab
- Part 2: Dose Escalation with Fractionated Dosing: RO7507062 (Experimental): Participants will receive RO7507062 as SC injection at the dose determined in Part 1, on Day 1 and as escalated doses on subsequent days.
  Interventions: Drug: RO7507062; Drug: Tocilizumab

INTERVENTIONS:
Drug: RO7507062 — RO7507062 solution for injection will be administered SC as specified in each treatment part (arm).
Drug: Tocilizumab — When applicable, tocilizumab solution for infusion will be administered intravenously at 8 milligram per kilogram (mg/kg) for participants >/= 30 kg or at 12 mg/kg for participants < 30 kg.
  Other Names: Actemra, RoActemra

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of RO7507062 in participants with systemic lupus erythematosus (SLE). The study will have 2 parts: Part 1 is a single ascending dose-finding (SAD) part and Part 2 is a dose escalation with fractionated dosing part.

DETAILED DESCRIPTION:
Tocilizumab is an additional investigational medicinal product (IMP), which may be used at the investigator's discretion when required in case of clinical presentation of cytokine release syndrome (CRS).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of SLE according to the 2019 European League Against Rheumatism (EULAR) or American College of Rheumatology (ACR) Classification Criteria at least 24 weeks prior to Screening and should have been treated for SLE according to standard clinical practice.
* Presence of anti-double stranded DNA (dsDNA), anti-Smith (Sm), anti-ribonucleoprotein (RNP) or anti-Sjögren's syndrome antigen A (SS-A) above the upper limit of normal (ULN); or, positive anti-nuclear antibody (ANA; ≥ 1:160).
* Active SLE disease, as demonstrated by the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) total score of ≥4 with at least 1 positive clinical item.
* For participants receiving oral corticosteroids (OCS), treatment with ≤ 20 milligram per day (mg/day) prednisone or equivalent, during Screening, at a dose that has been stable for at least 7 days prior to Day 1.
* For participants receiving conventional immunosuppressants (e.g., azathioprine, sulfasalazine, mycophenolate mofetil [≤ 3.0 grams per day], mycophenolic acid [≤ 3 grams per day], methotrexate [oral, SC, or intramuscular routes]), and calcineurin inhibitors [oral]), treatment should be at a stable dose for at least 6 weeks prior to Screening and during Screening and expected to remain stable during the study.

Exclusion Criteria:

* Active or unstable lupus-associated neuropsychiatric disease.
* Catastrophic or severe antiphospholipid syndrome within 12 months prior to Screening or during Screening.
* Presence of severe lupus-associated renal disease that is likely to require treatment with cyclophosphamide, B-cell-depleting therapies, other biologic or targeted therapies.
* Organ-threatening SLE manifestations (e.g., active myocarditis) considered to be severe by the Investigator.
* Severe active systemic autoimmune disease other than SLE.
* Active infection of any kind, excluding fungal infection of the nail beds.
* History of serious recurrent or chronic infection, especially; recurring, chronic infections specifically related to respiratory issues.
* Moderate or severe chronic obstructive pulmonary disease (COPD).
* History of progressive multifocal leukoencephalopathy (PML).
* History of macrophage-activation syndrome and/or hemophagocytic lymphohistiocytosis.
* History of cancer, including solid tumors, hematological malignancies, and carcinoma in situ, within the 5 years prior to the Screening visit (with the exception of basal cell carcinoma, non melanoma skin cancer, and cervical cancer in situ, if these have been adequately treated and are considered cured).
* Intolerance or contraindication to study therapies including history of severe allergic or anaphylactic reactions to monoclonal antibodies (mAbs) or known hypersensitivity to any component of the RO7507062 injection.
* History of infection with hepatitis B virus (HBV), or positive serology indicative of current or past HBV infection.
* Human immunodeficiency virus (HIV; positive HIV antibody test) and active hepatitis C virus (HCV) infection (detectable HCV ribonucleic acid [RNA]).
* Active cytomegalovirus (CMV) or Epstein-Barr virus (EBV) infection.
* Receipt of any anti- cluster of differentiation (CD)19 or anti-CD20 therapy such as blinatumomab, obinutuzumab, rituximab, ocrelizumab, or ofatumumab less than 6 months prior to screening or during screening.
* Receipt of Inhibitors of Janus kinase (JAK), Bruton tyrosine kinase, or tyrosine kinase 2 including baricitinib, tofacitinib, upadacitinib, filgotinib, ibrutinib, and fenebrutinib,or any investigational agent within 30 days prior to screening or during screening.
* Receipt of Cyclophosphamide or a biologic therapy such as, but not limited to, adalimumab, etanercept, golimumab, infliximab, belimumab,ustekinumab, anifrolumab, secukinumab, or atacicept, within 4 weeks prior to enrollment.
* Active tuberculosis or history of recurring or severe active tuberculosis, or a positive Interferon Gamma Release Assay (IGRA). Latent tuberculosis which has been treated prior to baseline is not exclusive.
* Receipt of an investigational therapy (except severe acute respiratory syndrome coronavirus 2 [SARS-CoV-2] vaccines) within 30 days or 5 drug-elimination half-lives (whichever is longer) prior to initiation of study treatment and during the study.
* Immunoglobulin (IgG) level of <6 gram per liter (g/L).
* Estimated glomerular filtration rate (eGFR) <45 milliliter per minute (mL/min)/1.73-meter square (m^2).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Dose Limiting Adverse Events (DLAEs) | Day 1 through Day 29
Part 2: Fractionated Dose Cohort: Number of Participants with DLAEs | Day 1 through to the end of the 28-day safety evaluation period
Number of Participants with Adverse Events (AEs) | Up to approximately 12 months
  Adverse events will be reported according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0), and CRS, will be graded based on the American Society for Transplantation and Cell Therapy (ASTCT) criteria.

SECONDARY OUTCOMES:
Serum Concentration of RO7507062 | Up to approximately 12 months
Time to Maximum Serum Concentration (Tmax) of RO7507062 | Up to approximately 12 months
Maximum Serum Concentration (Cmax) of RO7507062 | Up to approximately 12 months
Area Under the Serum Concentration Versus Time Curve Extrapolated to Infinity (AUCinf) of RO7507062 | Up to approximately 12 months
Area Under the Serum Concentration Versus Time Curve From Time Zero to the Last Measurable Concentration (AUClast) of RO7507062 | Up to approximately 12 months
Apparent Terminal Half-Life (T1/2) of RO7507062 | Up to approximately 12 months
Terminal Rate Constant (λz) of RO7507062 | Up to approximately 12 months
Apparent Volume of Distribution (Vz/F) of RO7507062 | Up to approximately 12 months
Apparent Total Body Clearance (CL/F) of RO7507062 | Up to approximately 12 months
Number of Participants with Anti-Drug Antibodies (ADAs) to RO7507062 | Up to approximately 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (24):
- Colombia (3):
  - Clinica De La Costa, Barranquilla
  - Hospital Pablo Tobon Uribe, Medellín
  - Oncomedica S.A., Montería
- France (2):
  - Hôpital Saint Eloi, Montpellier
  - Groupe Hospitalier Pitie-Salpetriere, Paris
- Germany (2):
  - Charité Research Organisation GmbH, Berlin
  - Universitätsklinikum Duesseldorf, Düsseldorf
- Hospital Umum Sarawak, Kuching, Malaysia
- Mexico (3):
  - CREA Hospital Mexico Americano, Guadalajara, Jalisco
  - Hospital Angeles De Lindavista, Mexico City, Mexico CITY (federal District)
  - Hospital General De Mexico, Mexico City, Mexico CITY (federal District)
- Centre For Human Drug Research, Leiden, Netherlands
- Clínica San Juan Bautista CSJB, Lima, Peru
- Poland (3):
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Późna
  - MICS Centrum Medyczne Damiana, Walbrzyska, Warsaw
  - Wojskowy Instytut Medyczny- Panstwowy Instytut Badawczy, Warsaw
- FARMOVS (Pty) Ltd, Bloemfontein, South Africa
- Spain (3):
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Taiwan (2):
  - Chung Shan Medical University Hospital, Taichung
  - Chang Gung Medical Foundation - Linkou, Taoyuan District
- Ramathibodi Hospital, Mahidol Uni, Bangkok, Thailand
- UCL Hospital NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No